CLINICAL TRIAL: NCT02340442
Title: Retinal Vessel Analysis in Low Risk and High Risk Pregnant Women
Brief Title: DVA Risk Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Harald, Zeisler, Prof. Dr., Medical University of Vienna
Other Study IDs: OPHT-060513
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pregnancy; High Risk Pregnancies
Keywords: arteriovenous ratio; retinal flicker stimulation; Dynamic vessel analyzer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Low risk group: 40 subjects: Healthy, pregnant women
  Interventions: Other: Obstetrical care parameters; Other: DVA measurements; Other: Fundus photographs
- High risk group: 40 pregnant women:
  * 20 Pregnant women with preeclampsia
  * 20 Obese pregnant women
  Interventions: Other: Obstetrical care parameters; Other: DVA measurements; Other: Fundus photographs
- Healthy control subjects: 40 subjects
  Interventions: Other: Obstetrical care parameters; Other: DVA measurements; Other: Fundus photographs

INTERVENTIONS:
Other: Obstetrical care parameters
Other: DVA measurements
Other: Fundus photographs

SUMMARY:
Maternal obesity, overweight and hypertensive disorders are among the most important risk factors for complications during pregnancy. Several lines of evidence indicate that overweight or obese women, as well as women with hypertensive disorders show increased risks of preterm birth before 32 weeks. However, an easy to determine, common reliable prognostic factor which allows for the early identifications of risk patients is still lacking. Recently, it has been reported that assessment of endothelial function may be a new promising tool for predicting the risk of adverse pregnancy outcome. As such evidence has been provided that endothelial dysfunction is prevalent among women with preeclampsia and is able to identify women at increased risk of preterm delivery and small-for-gestational-age (SGA) births. Several lines of evidence indicate that functional and structural changes of retinal vessels are altered in vascular related disease and may predict cardio-vascular events. Consequently, the current study seeks to investigate whether flicker induced vasodilatation, a well established parameter to test vascular function in-vivo is altered in women with low and high risk pregnancies when compared to a healthy control group. The data gained from this study may provide the basis for a larger longitudinal trial to assess whether vascular changes in the retina may predict the risk for complication during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years

  * Written informed consent
  * Pregnancy at screening
  * Normal ophthalmic findings, unless the investigator considers a finding clinically irrelevant.
  * Ametropy <= 3,5 Dpt.

For pregnant women with preeclampsia:

* Systolic BP ≥140 mmHg, or diastolic BP ≥90 mmHg on at least 2 occasions AND
* Proteinuria (≥300 mg/day) after 20 weeks of gestation in preeclampsia
* Pregnant at the time of confirming diagnosis of preeclampsia

For pregnant women with obesity:

• Pre-pregnancy BMI ≥30 as assessed from medical history

According to the WHO BMI classification:

* Underweight (less than 18.5)
* normal weight (18.5-24.9)
* overweight (25-29.9)
* obese class I (30 -34.9)
* obese class II (35-39.9)
* obese class III (40 or more) For non-pregnant control subjects

  * Age >18 years
  * Written informed consent
  * Not pregnant at screening
  * Normal ophthalmic and medical findings, unless the investigator considers a finding clinically irrelevant.
  * Ametropy <= 3,5 Dpt.

Exclusion Criteria:

* Diabetes mellitus type I or II
* Renal failure requiring dialysis
* Cirrhosis of liver
* Collagenosis
* Vasculitis
* Paraproteinaemia
* Alcohol abuse
* Amyloidosis
* Clinical signs of polyneuropathy
* Any other clinical finding, unless the clinical investigator considers a finding to be non clinically significant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited form the gynecology department and the department of clinical pharmacology
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
flicker-induced retinal vasodilatation | at inclusion, 3 Trimenon, post partum

SECONDARY OUTCOMES:
adverse pregnancy outcome | post partum

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Department of Clinical Pharmacology, Vienna, Vienna
  - Department of Gynecology, Vienna, Vienna